CLINICAL TRIAL: NCT05596721
Title: Effect of Azithromycin With ICS/LABA in Non-eosinophilic Chest Tightness Variant Asthma: a Multicentre Randomized Trial
Brief Title: Azithromycin Treatment for Non-eosinophilic Chest Tightness Variant Asthma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZNECTVA
Record Dates: First submitted 2022-10-25; First posted 2022-10-27 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Asthma; Chest Syndrome; Azithromycin; Effect of Drug
Keywords: non-eosinophilic; chest tightness variant asthma; azithromycin; asthma control
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Azithromycin + ICS/LABA (Experimental): Azithromycin: 500mg, po, 3 times per week for 12w ICS/LABA: Budesonide and Formoterol Fum arate Powder for Inhalation, 1 inhale, bid for 12w
  Interventions: Drug: Azithromycin; Drug: ICS/LABA
- ICS/LABA (Placebo Comparator): ICS/LABA: Budesonide and Formoterol Fum arate Powder for Inhalation, 1 inhale, bid for 12w
  Interventions: Drug: ICS/LABA

INTERVENTIONS:
Drug: Azithromycin — Treat patient with azithromycin for 12w.
  Arms: Azithromycin + ICS/LABA
Drug: ICS/LABA — Treat patient with ICS/LABA according to Global Initiative for Asthma (GINA) guideline.

SUMMARY:
Bronchial asthma (abbr. asthma) is one of common airway chronic inflammatory disease which usually threatens human health. Typical symptoms of asthma are recurrent wheezing, shortness of breath, chest tightness and cough, usually happened at night or in early morning. However, there are still some patients who persist only clinical manifestations of chest tightness, namely, chest tightness variant asthma (CTVA). This subgroup of asthma usually lacks asthma-specific clinical features, therefore, often misdiagnosed and lack of effective treatment for a long time. The investigators' previous studies have found that CTVA has eosinophilic and non-eosinophilic subtypes. These patients with non-eosinophilic CTVA (NE-CTVA) are not sensitive to ICS/LABA, which guidelines recommend. At present, the specific treatment plan for NE-CTVA is urgently needed to elucidate. Azithromycin has immunomodulatory and anti-inflammatory effects in addition to their antibacterial effects. Maintenance treatment with azithromycin has been proved to be effective in chronic neutrophilic airway diseases and severe asthma. However, there are no clinical studies to confirm the effectiveness of azithromycin in non-eosinophilic asthma, especially atypical asthma such as NE-CTVA. Now the investigators performed a national multi-center study to explore whether azithromycin improves asthma symptom control and improves quality of life in people with NE-CTVA. Finally, to find an optimal treatment for NE-CTVA.

DETAILED DESCRIPTION:
Bronchial asthma (abbr. asthma) is one of common airway chronic inflammatory disease which usually threatens human health. Typical symptoms of asthma are recurrent wheezing, shortness of breath, chest tightness and cough, usually happened at night or in early morning. However, there are still some patients who persist only clinical manifestations of chest tightness. Focus on this group of patients, the investigators proposed a subgroup of bronchial asthma, namely, chest tightness variant asthma (CTVA). This subgroup of asthma usually lacks asthma-specific clinical features such as wheezing, shortness of breath, wheezing, therefore, often misdiagnosed for a long time.

The investigators' previous studies have found that CTVA is like the clinical classification of common asthma and cough variant asthma (CVA), and there are also eosinophilic and non-eosinophilic subtypes in CTVA. These patients with non-eosinophilic CTVA (NE-CTVA) are not sensitive to ICS/LABA, which guidelines recommend, and have lower FeNO values than sensitive CTVAs. At present, the specific treatment plan for NE-CTVA is a special clinical asthma phenotype, and further clinical studies are urgently needed to elucidate.

Azithromycin has immunomodulatory and anti-inflammatory effects in addition to their antibacterial effects. Maintenance treatment with azithromycin has been proved to be effective in chronic neutrophilic airway diseases including chronic obstructive pulmonary disease, cystic fibrosis, bronchiectasis and diffuse panbronchiolitis. Whilst azithromycin is effective and recommended in current American Thoracic Society (ATS) / European Respiratory Society (ERS) and Global Initiative for Asthma (GINA) guidelines for selected persistently symptomatic adults with severe asthma. However, there are no clinical studies to confirm the effectiveness of azithromycin in non-eosinophilic asthma, especially atypical asthma such as NE-CTVA.

The investigators conduct a national multi-center, prospective randomized trial to test the hypothesis that azithromycin improves symptom control and improves quality of life in people with NE-CTVA. To this end, the recruited participants will be randomly divided into ICS/LABA + azithromycin group and ICS/LABA group. The treatment period is 12 weeks, and then to evaluate the revised-asthma control questionnaire (r-ACQ) score, asthma quality of life questionnaire (AQLQ) score, self-rating anxiety scale (SAS), self-rating depression scale (SDS), lung function, and numbers of emergency or hospitalization. Provide clinical evidence for the optimal treatment of NE-CTVA.

ELIGIBILITY:
Inclusion Criteria:

1. all subjects agreed to participate, understand the project, observe the use of drugs, agree to follow-up, and signed informed consent;
2. the age of more than 14 and less 80 years old, gender and ethnicity are not limited;
3. the duration time was more than 6 months,and chest tightness was the only complaint, without breathing, short of breath, chronic cough;
4. no wheezing;
5. a diagnosis of asthma supported by one or more other characteristics:

   * bronchial provocation test positive;
   * improvement in forced expiratory volume at one second (FEV1) of more than 12% and 200 ml after inhaled salbutamol;
   * variability in diurnal peak expiratory flow (PEF) of more than 10% for one day during one week.
6. blood eosinophils < 150/µl and FeNO < 20 ppb;
7. exclude the following diseases by the corresponding doctors: coronary heart disease, myocarditis, heart failure, GERD, neuromuscular disease, and mental disease.

Exclusion Criteria:

1. can not cooperate with related inspection or for other reasons;
2. patients with chronic obstructive pulmonary disease, interstitial pneumonia, active tuberculosis, community acquired pneumonia, lung cancer, bronchiectasis, cor pulmonale, pulmonary embolism, and accompanied with serious systematic disease (such as coronary heart disease, myocarditis, heart failure, gastroesophageal reflux disease, neuromuscular disease, etc);
3. history of chronic hepatic kidney or neurologic disorder;
4. history of drug abuse, alcohol abuse or anesthesia or with a history of mental illness (schizophrenia, obsessive-compulsive disorder, depression) and against personality, motivation, suspicious, or other emotional or mental issues that may affect participation in the study;
5. taking part in other drug clinical trial project, or drop out less than 3 months;
6. during pregnancy, lactation women;
7. obvious abnormal of High Resolution CT;
8. macrolide allergy;
9. received azithromycin treatment in the past 2 weeks;
10. hearing impairment or abnormally prolonged QTc interval.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
r-ACQ | Change from Baseline ACQ at 12 weeks
  Revised-asthma control questionnaire.

SECONDARY OUTCOMES:
FEV1 | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Perform pulmonary function tests of patients and record the forced expiratory volume in one second.
Airway responsiveness | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Perform pulmonary function tests of patients and record the PD20-FEV1.
PEF | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Perform pulmonary function tests of patients and record the peak expiratory flow.
AQLQ | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Asthma quality of life questionnaire.
SAS | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Self-rating Anxiety Scale.
SDS | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Self-rating Depression Scale.
Numbers of emergency or hospitalization | Change from Baseline at 4 weeks, 8 weeks, and 12 weeks
  Record the numbers of emergency or hospitalization because asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Huahao Shen, M.D., Study Chair — The Second Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (13):
- China (13):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital,Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Central Hospital of Shenyang Military, Shenyang, Liaoning
  - Xijing Hospital, Xi'an, Shaanxi
  - Qilu Hospital, Shandong University, Jinan, Shandong
  - Changhai Hospital, Second Military Medical University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang